CLINICAL TRIAL: NCT00507429
Title: A Phase II/III Study to Evaluate the Safety and Efficacy of Combretastatin A-4 Phosphate in Combination With Paclitaxel and Carboplatin in Comparison With Paclitaxel and Carboplatin Against Anaplastic Thyroid Carcinoma [FACT]
Brief Title: Study of Combretastatin and Paclitaxel/Carboplatin in the Treatment of Anaplastic Thyroid Cancer
Acronym: FACT
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low rate of subject accrual
Sponsor: Mateon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXC4T4-302
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-02

CONDITIONS: Anaplastic Thyroid Cancer
Keywords: thyroid neoplasms; thyroid cancer; thyroid carcinoma
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic; Thyroid Neoplasms | interventions — combretastatin; fosbretabulin; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: CA4P + Carboplatin + paclitaxel (Experimental): Six 21-day cycles: CA4P (60 mg/m2 on Days 1, 8, 15), carboplatin (AUC 6) + paclitaxel (200 mg/m2) on Day 2
  Interventions: Drug: CA4P
- Arm 2: Carboplatin + Paclitaxel (Active Comparator): Six 21-day cycles of Carboplatin (AUC 6) + paclitaxel (200 mg/m2) given on Day 1
  Interventions: Drug: paclitaxel; Drug: carboplatin

INTERVENTIONS:
Drug: CA4P — CA4P 60mg/m squared for Days 1, 8, 15 for 6 cycles
  Other Names: combretastatin; fosbretabulin; Zybrestat
  Arms: Arm 1: CA4P + Carboplatin + paclitaxel
Drug: paclitaxel — 200mg/m squared on Day 1
  Other Names: Taxol; Paxene
  Arms: Arm 2: Carboplatin + Paclitaxel
Drug: carboplatin — 6 AUC on Day 1 following paclitaxel
  Other Names: Paraplatin
  Arms: Arm 2: Carboplatin + Paclitaxel

SUMMARY:
The purpose of the study is to determine the safety and efficacy of combretastatin combined with paclitaxel and carboplatin in the treatment of anaplastic thyroid cancer (ATC).

DETAILED DESCRIPTION:
Anaplastic thyroid carcinoma (ATC) is a high-grade neoplasm, characterized by an aggressive clinical course with brief survival, and refractoriness to currently available local and systemic modalities of treatment. There is no standard therapy for ATC, and no randomized comparative trials have been known to be conducted in this disease. One potential strategy is to combine the anti-tumor activity of the vascular disrupting agent combretastatin with conventional cytotoxic agents. This study will compare the overall survival of ATC patients treated with the triplet combination of combretastatin, paclitaxel, and carboplatin compared with the doublet treatment of paclitaxel and carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Anaplastic thyroid carcinoma histologically or cytologically confirmed by a pathology review
* Refractory to or progressed during or after therapy, or relapsed within 6 months following initial combined modality therapy (usually including systemic chemotherapy and radiation) for regionally advanced disease
* Systemic therapy is limited to one chemotherapy regimen that is clearly administered contiguously, (i.e., in an uninterrupted primary therapeutic approach)
* Prior radiation: 3 weeks must have elapsed since radiation and disease must be present beyond radiation ports
* Minimum of 3 weeks must have elapsed from the time of last chemotherapy prior to the first dose of study drug
* Patients with bulky thyroid/neck masses and/or suspicion of airway obstruction must undergo screening (indirect and direct laryngoscopy) to ensure patency of the trachea/airway prior to study enrollment and treatment
* ECOG Performance Score less than or equal to 2
* Adequate bone marrow reserve as evidenced by absolute neutrophil count (ANC) greater than 1,500/microL, platelet count greater than 75,000/microL.
* Adequate renal function as evidenced by serum creatinine less than or equal to 2.0 mg/dL (less than 177 micromol/L)
* Adequate hepatic function as evidenced by serum total bilirubin less than 2X greater than the upper limit of normal (ULN) (less than3X ULN in patients with liver metastases), AST (aspartate aminotransferase)/ALT (alanine aminotransferase) less than or equal to 3X the ULN for the local reference lab (less than or equal to 5X the ULN for patients with liver metastases)
* No clinically important sequelae from any prior surgery or radiotherapy.

Exclusion Criteria:

* Tumors confined to the thyroid.
* Clinically evident brain metastasis, including symptomatic involvement, evidence of cerebral edema by CT or MRI, radiographic evidence of progression of brain metastasis since definitive therapy, or continued requirement for corticosteroids
* Patients who receive chemotherapy for metastatic disease after completion of a combined modality approach.
* History of malignancies other than ATC except curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or localized prostate cancer with a current PSA of less than 4.0 mg/dL or microg/L
* Known hypersensitivity to CA4P, paclitaxel or carboplatin, or any of their components
* Receiving concurrent investigational therapy or who have received investigational therapy for any indication within 28 days of the first scheduled day of dosing
* Greater than Grade 2 peripheral neuropathy
* History of prior cerebrovascular event, including transient ischemic attack
* Uncontrolled hypertension (blood pressure greater than 150/100 mm Hg despite medication)
* Symptomatic vascular disease (e.g. intermittent claudication)
* History of unstable angina pectoris pattern, myocardial infarction (including non-Q wave MI) within the past 6 months, or NYHA Class III and IV congestive heart failure
* History of torsade de pointes
* Bradycardia (less than 60 b/m), heart block (excluding 1st degree block, being PR interval prolongation only), and congenital long QT syndrome
* Any ventricular arrhythmias, or new ST segment elevation or depression or Q wave on ECG
* Ejection fractions less than normal (i.e. less than 45%)
* QTc prolongation greater than 450 ms
* Requirement of any drugs known to prolong the QTc interval, including anti-arrhythmic medications
* Potassium concentrations below 4.0 mEq/dL and magnesium concentrations below 1.8 mg/dL despite being on an electrolyte supplement
* Requirement of any drugs known to prolong the QTc interval
* History of solid organ transplant or bone marrow transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-08; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A. Sosa, MD, FACS, Principal Investigator — Yale University School of Medicine, New Haven, CT
Locations (41):
- United States (10):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale University, School of Medicine, New Haven, Connecticut
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Care Center at John Hopkins, Baltimore, Maryland
  - University of Minnesota Otolaryngology Department, Minneapolis, Minnesota
  - Ireland Cancer Center/Division od Hematology, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - West Virginia University, Morgantown, West Virginia
- Belarus National Medical University, Minsk, Belarus
- Bulgaria (3):
  - Regional Oncology Dispensary with Inpatient Sector, Plodiv
  - Specialized Hospital for Active Treatment of Oncology, Sofia
  - Universtiy Multiprofile Hospital, ISUI, Clinic of Oncotherapy, Sofia
- University Hospital, Cairo, Cairo, Egypt
- India (8):
  - Mediciti Hospital, Hyderabaad, Andhra Pradesh
  - Kidwai Memorial Hospital, Bangalore, Karnataka
  - Shirdi Sai Baba Cancer Hospital, Manipal, Karnataka
  - Tata Memorial Centre, Mumbai, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Apollo Cancer Institute, New Delhi, National Capital Territory of Delhi
  - Christian Medial College, Vellore, Tamil Nadu
- Telaviv Sourasky Medical Center, Head and Neck Service Division of Oncology, Tel Aviv, Israel
- Italy (4):
  - Lo Studio E la Cura, Milan
  - INT Napoli Fondazione Pascale, Napoli
  - Istituto Oncologico Veneto (IOV) - IRCCS, Padua
  - Azienda Ospedaliero - Universitaria Pisana, Pisa
- Poland (2):
  - Zaklad Medyczny Nuklearnej i Endykrynologii, Gliwice
  - Klinika Nowotworow Glowy i Szyji, Warsaw
- Romania (5):
  - Institutul Oncologic, Cluj-Napoca
  - SC Meditech SRL, Craiova
  - Centr of Medical Oncology, Iași
  - Clinical County Hospital Sibiu, Sibiu
  - Emergency Clinical County Hospital "Sf. loan cel Nou", Suceava
- City Clinical Oncology Dispensary, Saint Petersburg, Russia
- Ukraine (2):
  - Ukrainian Academy of Medical Science, Lomonosova 33/43, Kiev
  - Regional Clinical Oncology Dispensary, Lviv
- United Kingdom (3):
  - Beatson Oncology Centre, Gartnavel General Hospital, Glasgow, Scotland
  - Royal Marsden Hospital and Institute of Cancer Research, London
  - Southampton Hospital Oncology Centre, Southampton

REFERENCES:
- [Background] Yeung SC, She M, Yang H, Pan J, Sun L, Chaplin D. Combination chemotherapy including combretastatin A4 phosphate and paclitaxel is effective against anaplastic thyroid cancer in a nude mouse xenograft model. J Clin Endocrinol Metab. 2007 Aug;92(8):2902-9. doi: 10.1210/jc.2007-0027. Epub 2007 Jun 5. PMID 17550961
- [Background] Patel KN, Shaha AR. Poorly differentiated and anaplastic thyroid cancer. Cancer Control. 2006 Apr;13(2):119-28. doi: 10.1177/107327480601300206. PMID 16735986
- [Background] Ain KB. Anaplastic thyroid carcinoma: behavior, biology, and therapeutic approaches. Thyroid. 1998 Aug;8(8):715-26. doi: 10.1089/thy.1998.8.715. PMID 9737368
- [Background] De Crevoisier R, Baudin E, Bachelot A, Leboulleux S, Travagli JP, Caillou B, Schlumberger M. Combined treatment of anaplastic thyroid carcinoma with surgery, chemotherapy, and hyperfractionated accelerated external radiotherapy. Int J Radiat Oncol Biol Phys. 2004 Nov 15;60(4):1137-43. doi: 10.1016/j.ijrobp.2004.05.032. PMID 15519785
- [Background] Siemann DW, Chaplin DJ, Horsman MR. Vascular-targeting therapies for treatment of malignant disease. Cancer. 2004 Jun 15;100(12):2491-9. doi: 10.1002/cncr.20299. PMID 15197790
- [Background] Horsman MR, Siemann DW. Pathophysiologic effects of vascular-targeting agents and the implications for combination with conventional therapies. Cancer Res. 2006 Dec 15;66(24):11520-39. doi: 10.1158/0008-5472.CAN-06-2848. PMID 17178843
- [Background] Cooney MM, Savvides P, Agarwala SS, Wang D, Flick S, Bergant S, Bhatka S,Fu P, Subbiah V, Lavertu P, Ortiz J, and Remick S. Phase II study of combretastatin A4 phosphate (CA4P) in patients with advanced anaplastic thyroid carcinoma. J Clinical Oncology, 2006 Vol. 24, 5580.
- [Derived] Giri P, Batra PJ, Kumari A, Hura N, Adhikary R, Acharya A, Guchhait SK, Panda D. Development of QTMP: A promising anticancer agent through NP-Privileged Motif-Driven structural modulation. Bioorg Med Chem. 2023 Nov 15;95:117489. doi: 10.1016/j.bmc.2023.117489. Epub 2023 Oct 5. PMID 37816266
- See also: Link to Thyroid Cancer Survivors website — http://www.thyca.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study truncated from 180 to 80 subjects. Subjects were enrolled from August 2007 through March 2010 at 40 worldwide, academic and local-regional clinical sites.
Pre-assignment Details: During screening, the diagnosis of anaplastic thyroid cancer was centrally confirmed often leading to enrollment and randomization delays.
Groups:
- Arm 1, Active: CA4P + Carboplatin + Paclitaxel: Randomized 2:1 to receive six 21-day cycles of CA4P (60mg/m2)on days 1, 8, 15 + carboplatin (AUC 6) + paclitaxel (200 mg/m2) on Day 2. Subjects without progressive disease may continue maintenance CA4P infusions until progressive disease, then followed monthly for survival.
- Arm 2, Control: Carboplatin + Paclitaxel: On Day 2 of six 21-cycles subjects received Carboplatin (AUC 6) + paclitaxel (200 mg/m2). Subjects without progressive disease were followed monthly for survival.
Period: Treatment Phase
Arm/Group | Arm 1, Active: CA4P + Carboplatin + Paclitaxel | Arm 2, Control: Carboplatin + Paclitaxel
Started | 55 (Randomized) | 25 (Randomized)
Completed | 18 | 7
Not Completed | 37 | 18
Not completed — Disease Progression | 12 | 5
Not completed — Adverse Event | 12 | 5
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Physician Decision | 4 | 2
Not completed — Other | 6 | 3
Period: Maintenance Phase
Arm/Group | Arm 1, Active: CA4P + Carboplatin + Paclitaxel | Arm 2, Control: Carboplatin + Paclitaxel
Started | 16 (2 subjects did not enter maintenance: 1/18 progressive disease; 1/18 lost to follow-up.) | 0 (Control arm subjects followed for survival only; not enrolled in Maintenance period)
Completed | 2 (14 subjects were withdrawn due to progressive disease, 2 subjects continued beyond data cut-off) | 0
Not Completed | 14 | 0
Not completed — Progressive Disease | 14 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1, Active: CA4P + Carboplatin + Paclitaxel | Arm 2, Control: Carboplatin + Paclitaxel | Total
Number analyzed (Participants) | 55 | 25 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 14 | 43
  >=65 years | 26 | 11 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (10.72) | 61.2 (10.54) | 61.4 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 43
  Male | 30 | 7 | 37
Region of Enrollment [Number; unit: participants]
  Belarus | 1 | 1 | 2
  United States | 20 | 5 | 25
  Poland | 5 | 1 | 6
  Ukraine | 1 | 1 | 2
  Romania | 1 | 0 | 1
  Russian Federation | 2 | 1 | 3
  Bulgaria | 3 | 0 | 3
  Israel | 2 | 1 | 3
  Italy | 13 | 8 | 21
  United Kingdom | 2 | 1 | 3
  India | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: From randomization to date last known alive
Population: All randomized subjects (the Intent-to-treat population) included in the analysis
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm 1, Active: CA4P + Carboplatin + Paclitaxel: Six 21-day cycles of CA4P (60 mg/m2) on days 1, 8, 15, carboplatin (AUC 6) and paclitaxel (200 mg/m2) on Day 2
- Arm 2, Comparator: Carboplatin + Paclitaxel: Six 21-day cycles of carboplatin (AUC 6) and paclitaxel (200 mg/m2) on Day 1
Arm/Group | Arm 1, Active: CA4P + Carboplatin + Paclitaxel | Arm 2, Comparator: Carboplatin + Paclitaxel
Number analyzed (Participants) | 55 | 25
months | 5.2 [3.1 to 9.0] | 4.0 [2.8 to 6.2]
Statistical Analysis 1: Comparison: Arm 1, Active: CA4P + Carboplatin + Paclitaxel vs Arm 2, Comparator: Carboplatin + Paclitaxel; Test type: Superiority or Other; p = 0.223, Log Rank

2. Secondary Outcome: To Determine Progression Free Survival
Time Frame: from randomization through end of study visit
Reporting Status: Not Posted

3. Secondary Outcome: To Determine Percentage of 1 Year Survival
Time Frame: from randomization through end of study visit
Population: Intent to treat
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1, Active: CA4P + Carboplatin + Paclitaxel | Arm 2, Control: Carboplatin + Paclitaxel
Number analyzed (Participants) | 55 | 25
percentage of participants | 26 | 9

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 2 years, 6 months. All serious adverse events were reported, regardless of relatedness. Adverse events occurring at a frequency of >/= 5% in either arm are reported, regardless of relatedness.
Description: The median duration of overall follow-up was 4.5 mos, with a range of 0.1 to 35.5 mos. The median follow-up for Arm 1 subjects was 5.1 mos compared to 3.9 mos for Arm 2 subjects. Median follow-up for the study drug treatment periods (exposure to study drugs) was 2.9 mos (range = 0.1-22.1 mos) for Arm 1 versus 2.8 mos (range 0.2-6.9 mos) Arm 2.
Arm/Group | Arm 1, Active: CA4P + Carboplatin + Paclitaxel | Arm 2, Comparator: Carboplatin + Paclitaxel
Serious Adverse Events (participants affected / at risk) | 21/51 | 5/24
Other Adverse Events (participants affected / at risk) | 50/51 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1, Active: CA4P + Carboplatin + Paclitaxel (N=51) | Arm 2, Comparator: Carboplatin + Paclitaxel (N=24)
Anemia (Blood and lymphatic system disorders) | 1 | 2
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis (Infections and infestations) | 5 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Edema peripheral (General disorders) | 1 | 0
Esophageal fistual (Gastrointestinal disorders) | 1 | 0
Esophageal obstruction (Gastrointestinal disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxic encephalopathy (Nervous system disorders) | 0 | 1
Intestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Necrosis (General disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Obstructive Airways Disorders (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Performance status decreased (General disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonay embolism (Reproductive system and breast disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Tumor hemorrhage (Blood and lymphatic system disorders) | 2 | 0
Tumor pain (General disorders) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1, Active: CA4P + Carboplatin + Paclitaxel (N=51) | Arm 2, Comparator: Carboplatin + Paclitaxel (N=24)
Abdominal pain (Gastrointestinal disorders) | 6 | 2
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0
Alanine transferase increased (Investigations) | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 3
Anemia (Blood and lymphatic system disorders) | 20 | 12
Anorexia (Metabolism and nutrition disorders) | 9 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 0
Asthenia (General disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 0
Blood thyroid stimulating hormone increased (Investigations) | 4 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Cachexia (Metabolism and nutrition disorders) | 4 | 0
Cellulitis (Infections and infestations) | 3 | 0
Chills (General disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 12 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Diarrhea (Gastrointestinal disorders) | 15 | 4
Disease Progression (General disorders) | 7 | 1
Dizziness (Nervous system disorders) | 4 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 0
Dysgeusia (Nervous system disorders) | 4 | 1
Dyspea (Respiratory, thoracic and mediastinal disorders) | 15 | 4
Dysphagia (Gastrointestinal disorders) | 15 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Electrocardiogram QT prolonged (Investigations) | 8 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 0
Fatigue (General disorders) | 18 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
Flushing (Vascular disorders) | 6 | 0
Headache (Nervous system disorders) | 14 | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Hypercholesterolemia (Metabolism and nutrition disorders) | 4 | 0
Hyperglycemia (Musculoskeletal and connective tissue disorders) | 4 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 0
Hypertension (Vascular disorders) | 18 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 9 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 7 | 1
Hyponatremia (Metabolism and nutrition disorders) | 4 | 1
Hypotension (Vascular disorders) | 6 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 21 | 2
Lymphopenia (Blood and lymphatic system disorders) | 5 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 2
Nausea (Gastrointestinal disorders) | 15 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 11 | 3
Neuropathy peripheral (Nervous system disorders) | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 30 | 7
Non-cardiac chest pain (General disorders) | 4 | 0
Obstructive airway disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Oedema peripheral (General disorders) | 5 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 2
Paraesthesia (Nervous system disorders) | 6 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 0
Pyrexia (General disorders) | 14 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Sinus tachycardia (Cardiac disorders) | 8 | 2
Tachycardia (Cardiac disorders) | 4 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 2
Tremor (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Upper respiratory infection (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 4 | 1
Vomiting (Gastrointestinal disorders) | 13 | 7
Weight decreased (Investigations) | 6 | 0

LIMITATIONS AND CAVEATS:
The study was to enroll 180 subjects. Enrollment was terminated early due to low accrual rate. Eighty subjects were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No